CLINICAL TRIAL: NCT06433037
Title: Gut-brain Health Effects of PREbiotics in Older Adults With Suspected COgnitive DEcline: The PRECODE Study
Brief Title: Gut-brain Health Effects of PREbiotics in Older Adults With Suspected COgnitive DEcline
Acronym: PRECODE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Sensus BV (Unknown); Cosun Nutrition Center (Unknown); Roquette Frères (Unknown); Oceanium Ltd. (Unknown); Technical University of Eindhoven (TU/e) (Unknown)
Responsible Party: Principal Investigator, Yannick Vermeiren, Assistant Professor in Nutrition, Brain and Cognitive Aging, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NL85910.091.23
Record Dates: First submitted 2024-05-17; First posted 2024-05-29 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Subjective Cognitive Decline
Keywords: gut-brain axis; working memory; gut health; dietary fibres; prebiotics

STUDY DESIGN:
Intervention Model Description: Randomised, double-blinded, placebo-controlled intervention study with parallel design and four arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Maltodextrin (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Chicory inulin (Experimental)
  Interventions: Dietary Supplement: Chicory inulin
- Resistant dextrin (Experimental)
  Interventions: Dietary Supplement: Resistant dextrin
- Seaweed polysaccharide (Experimental)
  Interventions: Dietary Supplement: Seaweed polysaccharide

INTERVENTIONS:
Dietary Supplement: Chicory inulin — Chicory inulin (12g/day) divided over two dosages (6g per dose)
  Arms: Chicory inulin
Dietary Supplement: Resistant dextrin — Resistant dextrin (14g/day) divided over two dosages (7g per dose)
  Arms: Resistant dextrin
Dietary Supplement: Seaweed polysaccharide — Seaweed polysaccharide (1g/day) divided over two dosages (0.5g per dose). Additionally contains 7g/day of placebo as a volumetric and isocaloric filler.
  Arms: Seaweed polysaccharide
Dietary Supplement: Placebo — Maltodextrin (7g/day) will be provided in two divided doses (3.5g per dose)
  Arms: Maltodextrin

SUMMARY:
As people around the world are living longer, the number of individuals with dementia, particularly Alzheimer's disease (AD), is expected to triple by 2050. There's growing evidence suggesting that our gut health might play a role in the prevention of dementia. The connection between our gut and brain, known as the gut-brain axis, is becoming an important area of study. Research in animals has shown that different types of dietary fibre can improve gut health, brain function, mood, blood sugar level and the immune system and may even prevent certain harmful brain changes seen in Alzheimer's disease. Subjective Cognitive Decline (SCD) is a condition where individuals notice a decline in their mental abilities, and it can be an early sign of Alzheimer's disease.

The goal of this clinical trial is to learn if dietary fibres can improve gut and brain health in older individuals, between the ages of 60 and 79 years, who notice problems in their mental abilities, and meet the criteria of SCD. Three different dietary fibres will be given, and researchers will compare three different fibres to a placebo product to see if there is a difference between the fibres and the placebo.

The main questions it aims to answer are:

1. Does dietary fibre improve working memory?
2. Does dietary fibre improve other markers of brain function?
3. Does dietary fibre improve gut health?
4. Does dietary fibre improve the immune system and blood glucose levels?
5. Does dietary fibre improve mood?

Participants will:

* Consume dietary fibres twice a day, mixed in water, tea or coffee, for a period of 26 weeks
* Have two functional MRI scans, and three additional study visits, where blood, urine and feces will be collected
* Undergo a number of neuropsychological tests, aimed at evaluating brain function
* Fill out questionnaires on their general health, mood, dietary habits, gut health
* Wear smartwatches for one week, at the beginning and the end of the study

DETAILED DESCRIPTION:
Rationale: Due to the greying of society, a triplication of the number of people with dementia worldwide, with Alzheimer's disease (AD) as the commonest form, is expected by 2050. Compelling evidence points towards a crucial role of intestinal health as one potential etiological modifier of dementia, with the (microbiota) gut-brain axis (MGBA) receiving increasing attention. A number of preclinical studies have demonstrated benefit of various sources of dietary fibre for their capacity to improve gut health, cognitive functioning, general mood, glycaemia, immunogenicity, and, to inhibit tau phosphorylation, the latter which is a hallmark in AD brain. Subjective cognitive decline (SCD) lies on the continuum of AD, and subjects with this condition are at increased risk of further conversion to mild cognitive impairment (MCI) or AD. Currently, no cure is available for AD. Various symptomatic and a few disease-modifying treatments are available, but these treatments only have very limited or mild clinical effects and are often accompanied by severe side effects. Clinical follow-up studies to evaluate the effect of dietary fibre in older adults with suspected cognitive decline are required, but are still lacking to date.

Objective: The primary objective of this study is to investigate the effect of 26 weeks of supplementation with three different dietary fibres (chicory inulin, resistant dextrin, and seaweed polysaccharide) compared to a placebo (maltodextrin) on microbiota gut-brain health effects in older adults (aged 60-79) with Subjective Cognitive Decline Plus (SCD+) by assessing changes in brain function and working memory by blood oxygen level dependant (BOLD) signal activity and task accuracy during n-back task functional magnetic resonance imaging (fMRI) assessment.

The secondary objectives are to investigate the effects of 26 weeks of supplementation with dietary fibre (chicory inulin, resistant dextrin, and, seaweed polysaccharide) compared to placebo (maltodextrin) in older adults on the following parameters related to potential gut-brain pathways:

1. neuropsychological test battery scoring,
2. other relevant brain health parameters,
3. relevant intestinal health parameters, and
4. immune and metabolic parameters.

Study population: 164 older adults (60-79 years) with SCD+.

Study design implementation:

Participants will undergo assessments at baseline (T0), mid-study (T1/2, after 13 weeks) and at study end (T1, after 26 weeks. Each participant will have five study visits in total: two at T0, one at T1/2 and two at T1.

At each of the timepoints the following will be collected/performed at WUR: Sample collection (blood, urine (omitted in week 13), faeces); general cognitive assessments (see NTB; Cognitive Failure Questionnaire (CFQ) (baseline and end only), GDS-15, GAD-7); general physiological measures (blood pressure, BMI, grip-strength); dietary assessment (MIND-adjusted Eetscore, FFQ). At ZGV working memory will be evaluated using BOLD fMRI signalling and task accuracy using an n-back task paradigm. Additionally, high-resolution T1- and T2-weighted anatomical images of main regions of interest (hippocampi, (pre)frontal-, and temporal cortices) will be acquired.

For two periods of one week, corresponding with the baseline and week 26 visits, participants will wear smartwatches. These watches will be worn continuously and data will be gathered regarding cardiovascular functioning (heart rate), physical activity and mood (push messages).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Fluency in Dutch (speaking, reading, writing)
3. Age between 60-79 years (at screening)
4. Subjective cognitive decline plus (SCD+), (criteria of Jessen et al.):

4.1 Self-reported worsening of memory; 4.2 Indication of repetitive concerns (worries) associated with SCD; 4.3 With at least one of the following two features present: (i) onset of SCD within the last 5 years; (ii) age at onset ≥60 years of age;

5. Presence of at least 2 self-reported risk factors for cognitive decline (based on LIBRA criteria): (i) Diabetes mellitus type II (ii) High cholesterol (iii) Hypertension (iv) High BMI (v) Heart disease (vi) Unhealthy diet (lower regular adherence to Mediterranean diet components such as fish, vegetables, olive oil, pasta and red wine)

Exclusion Criteria:

1. Current participation in other intervention trials
2. Technologically illiterate (complete incompetence in working with computers, apps, online questionnaires, smartwatches etc.)
3. No internet access from home
4. Clinical diagnosis of ≥1 of the following:

   * Neurological pathology (e.g. MCI, dementia, multiple sclerosis, Parkinson's disease, epilepsy);
   * Current malignant disease(s), with or without treatment;
   * Current psychiatric disorder(s) (e.g. major depressive disorder, bipolar disorder, schizophrenia, anxiety, psychosis, PTSD);
   * Symptomatic/decompensated cardiovascular disease (e.g. stroke, angina pectoris, heart failure, recent myocardial infarction);
   * Severe visual impairment or blindness
   * Hearing or communicative impairment.
   * Gastrointestinal tract disorder such as irritable bowel syndrome or inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis).
5. Current or recent (<6 weeks) use of prebiotic, probiotic, or dietary fibre supplement that may modulate the microbiota, or unwilling to stop the use of supplements during the study
6. Current or recent (<6 weeks) of algae/phytoplankton supplements such as spirulina or chlorella, or unwilling to stop the use of supplements during the study
7. Use of psychotropic medication (anti-depressants, anti-psychotics)
8. Use of antibiotics in the 3 months before starting the study or planned use during the study
9. Being an employee of the Human Nutrition and Health Division of Wageningen University.
10. Significant cognitive impairment assessed using the Modified Telephone Interview for Cognitive Status battery (TICS-m score <23)
11. Request to have Apo-E genotype result disclosed
12. Allergies to fish or shellfish
13. Having a contra-indication to MRI scanning including:

    * Ferromagnetic implants:

      * Active implantable medical devices such as: insulin pump / medicine pump / neurostimulator; pacemaker / defibrillator;
      * Other passive implants such as: punctured port-a-cath; synthetic heart valve
    * Intra-orbital or intra-ocular metallic fragments
    * Claustrophobia

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Effect on working memory during n-back task fMRI | Measured at baseline and week 26
  Effects on working memory will be assessed by blood-oxygen level dependant (BOLD) signal activity during 2-back task performed during fMRI scanning
Effect on working memory performance during n-back task fMRI | Measured at baseline and week 26
  Effects on working memory performance will be assessed by task accuracy during 2-back task performed during fMRI scanning

SECONDARY OUTCOMES:
Effect on cognitive functioning as measured by a neuropsychological test battery | Measured at baseline, week 13 and week 26
  Effect on z-scoring of cognitive domains- episodic memory, executive function and working memory as measured by Cognitive Function Composite test battery
Effect on ADAS-Cog Word Recall cognitive assessment (episodic memory) | Measured at baseline, week 13 and week 26
  Mean number of correct responses across three trials; Score 0 to 10. Higher score indicates better outcome.
Effect on ADAS-Cog Word Recognition cognitive assessment (episodic memory) | Measured at baseline, week 13 and week 26
  Mean number of correct responses across three trials. Score 0 to 12. Higher score indicates better outcome.
Effect on Digit Symbol Substitution Test cognitive assessment (executive function) | Measured at baseline, week 13 and week 26
  Amount of symbols correctly substituted. Score 0 - 90. Higher score indicates better outcome
Effect on Digit Span Backward Task cognitive assessment (working memory) | Measured at baseline, week 13 and week 26
  Longest span of digits correctly recalled. Score 2-8. Higher score indicates better outcome
Effect on Category Fluency Test cognitive assessment (executive function) | Measured at baseline, week 13 and week 26
  Number of uniquely named items from category within 60 seconds. Higher score indicates better outcome
Effect on ADAS-Cog Orientation cognitive assessment (episodic memory) | Measured at baseline, week 13 and week 26
  The number of correct responses on orientation. Score 0 to 8. Higher score indicates better outcome
Effect on tryptophan metabolites | Measured at baseline and week 26
  Tryptophan related neurotransmitters and metabolites (plasma)
Effect on amyloid-beta (Aβ) biomarker | Measured at baseline and week 26
  Aβ1-42/Aβ1-40 ratio (plasma)
Effect on neuroplasticity | Measured at baseline and week 26
  Brain-derived neurotrophic factor (BDNF) levels (serum)
Effect on brain regions of interest | Measured at baseline and week 26
  Structural MRI with T1- and T2-weighted anatomical images of regions of interest (hippocampi, (pre)frontal-and temporal cortices)
Effect on hypothalamic-pituitary adrenal axis | Measured at baseline and week 26
  Cortisol levels (serum)
Effect on intestinal barrier integrity | Measured at baseline, week 13 and week 26
  Assay-based panel of intestinal barrier integrity markers measured in blood
Effect on intestinal inflammation | Measured at baseline, week 13 and week 26
  Assay-based panel of intestinal inflammatory markers measured in faeces
Effect on gastrointestinal transit time | Measured at baseline, week 13 and week 26
  Gut transit time measured by blue muffin consumption and appearance of blue colour in faeces
Effect on gastrointestinal symptoms | Measured at baseline, week 13 and week 26
  Self-rated gastrointestinal symptoms as measured by the Gastrointestinal Symptom Rating Scale (GSRS) questionnaire
Effect on self-reported stool consistency | Measured at baseline, week 13 and week 26
  Effect on stool consistency as measured by Bristol Stool Scale (BSS)
Effect on stool consistency | Measured at baseline, week 13 and week 26
  Effect on stool consistency as measured by faecal water content
Effect on qualitative faecal microbiota composition | Measured at baseline, week 13 and week 26
  Qualitative faecal microbiota composition as measured by 16s rRNA sequencing
Effect on quantitative faecal microbiota composition | Measured at baseline, week 13 and week 26
  Quantitative faecal microbiota composition as measured by digital droplet PCR
Effect on faecal metabolites | Measured at baseline, week 13 and week 26
  Faecal short-chain fatty acids (acetic acid, propionic acid, butyric acid, valeric acid, hexanoic acid, heptanoic acid) and branched-chain fatty acids (isobutyric acid, isovaleric acid, 4-methyl valeric acid) as measured by gas chromatography-flame ionization detection (GC-FID)
Effect on faecal pH | Measured at baseline, week 13 and week 26
  Faecal pH measurement
Effect on immune parameters | Measured at baseline, week 13 and week 26
  Inflammatory cytokine panel measured in blood
Effect on glucose homeostasis | Measured at baseline, week 13 and week 26
  Assay-based panel of markers to evaluate glucose homestasis in blood
Effect on lipid profile | Measured at baseline, week 13 and week 26
  Assay-based panel of markers to analyse lipid profile in blood

OTHER OUTCOMES:
Effect on heart rate | Measured at baseline and week 26
  Heart rate as determined by wearable Samsung Active 2.0 Smartwatches
Effect on physical activity | Measured at baseline and week 26
  Physical activity (pedometer) as determined by wearable Samsung Active 2.0 Smartwatches
Effect on BMI | Measured at baseline, week 13 and week 26
  Measured in kg/m^2
Effect on blood pressure | Measured at baseline, week 13 and week 26
  Systolic and diastolic blood pressure as measured by sphygmomanometer
Effect on mood as measured by Samsung Active 2.0 Smartwatches | Measured at baseline, week 13 and week 26
  Mood determined by push notifications (sad, stressed, neutral, happy, or angry) as determined by wearable Samsung Active 2.0 Smartwatches
Effect on mood as determined by GDS-15 questionnaire | Measured at baseline, week 13 and week 26
  Self-reported depressive symptoms by Geriatric Depression Scale-15 (GDS-15) questionnaire
Effect on mood as determined by GAD-7 questionnaire | Measured at baseline, week 13 and week 26
  Self-reported anxiety symptoms by Generalised Anxiety Disorder-7 (GAD-7) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PRECODE study Wageningen University — http://www.wur.nl/en/research-results/research-institutes/food-biobased-research/show-fbr/gut-brain-health-effects-of-prebiotics-in-older-adults-with-suspected-cognitive-decline-the-precode-study.htm